CLINICAL TRIAL: NCT01265056
Title: The Effect of Neurontin on Pain Management in the Acutely Burned Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucy A Wibbenmeyer (Other)
Responsible Party: Sponsor-Investigator, Lucy A Wibbenmeyer, Associate Clinical Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200909736
Record Dates: First submitted 2010-12-20; First posted 2010-12-22 (Estimated); Results first posted 2013-02-26 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Pain; Burn Injury
MeSH Terms: conditions — Pain; Burns | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participant, Care Provider and Investigator are all masked.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar Pill (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Gabapentin (Experimental): Gabapentin
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — On Study day 1: 1200mg (single dose).
  Study day 2,3: 300mg TID, 900mg daily.
  Study day 4-7: 600mg TID 1800mg* daily.
  Study day 8-11: 800mg TID 2400mg* daily [Optional increase to 2400 if pain scores are still 4 on NRS]
  Study day 11: 1200mg TID 3600mg* daily [Optional increase to 3600 if pain scores are still >4 on NRS]
  * May revert back to prior dose if adverse symptoms occur and are thought to be drug related. Up titration then will be preformed in 48 hours following deexcalation.
  Other Names: Neurontin
  Arms: Gabapentin
Drug: Placebo — Sugar Pill is administered similar to the protocol used for the investigational drug.
  Arms: Sugar Pill

SUMMARY:
Burn patients have extreme pain. Opioids are the main agents used for analgesia. We therefore propose a single center study to fruther assess the efficacy of neuropathic agents in controlling the pain associated with acute thermal injury.

DETAILED DESCRIPTION:
The study was conducted in a 16-bed American Burn Association certified burn unit. Patients age >18 years old, with at least a 5% burn injury and an expected length of stay (LOS) of 48 hours, were approached for enrollment in this prospective, placebo controlled randomized study. Patients who were pregnant, lactating, prisoners or who had renal insufficiency were excluded. After consent, patients were assigned to either placebo or Gp by random numbers generated in Microsoft Excel (2010). Both the drug and the placebo were over-encapsulated to appear identical. The placebo pills contained starch. The research clinical pharmacist was the only unblinded staff member and did not participate in clinical care of the patients.

Following randomization, patients received a loading dose of study drug on day one and began three times a day (TID) dosing per the dose escalation schedule the following day. At discharge, patients were given a three day taper per the dose de-escalation schedule Patients were assessed for completion of psychosocial adjustment (Brief Symptom Inventory, BSI, and Sickness Inventory Profile, SIP) at their first clinic visit.

Agents used for pain control included: acetaminophen, non-steroidal anti-inflammatories, morphine instantaneous release and morphine extended release. In the case of allergies or ineffectiveness, other agents were occasionally used. Short acting morphine was ordered every two hours prn and hydromorphone was ordered every four hours as needed. All were converted to morphine equivalents.

The study was powered to detect a 22% difference in opioid consumption between the two groups based on the work by Cuignet et al. It was estimated that a total of 50 patients were needed to achieve an alpha of 0.05 and a beta of 0.80 to detect the difference in the primary endpoint.

For statistical purposes, conversion tables were used to convert all opioid medications into morphine equivalents with 1 morphine equivalents (ME)=30mg oral morphine. The primary outcome variable (morphine consumption) were adjusted for days past injury. The BSI and SIP scales were scored according to study directions.

Both an intention to treat and actual treatment analysis were performed using Stata 11.2 for Windows (Stata Corp. College Station, Texas, U.S.A.). Continuous variables between groups were analyzed with the students T test. Categorical variables were analyzed with the Chi Square test or Fischer Exact Test where appropriate. A random effects model adjusting for confounders was used to assess the effect of treatment on the outcome measures. The study was approved by the University's Institutional Review Board and was registered with the clinical trials association (200909736).

ELIGIBILITY:
Inclusion Criteria:

* All admitted patients with LOS expected to be > 48 hours (usually burn injury > 5%)
* > 18 years of age
* Thermal injury to skin

Exclusion Criteria:

* Prisoners
* Pregnant or nursing women
* Children <18 years of age
* Frostbite or non thermal injury to skin
* Renal insuffiency (creatinine clearance < 60mL/min) or failure (on renal replacement)
* Expected length of stay < 48 hours (this usually includes burn <5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Wibbenmeyer, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Burn Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers can contact me (lucy-wibbenmeyer@uiowa.edu) for study protocol or statistical plan.
Supporting Information: Study Protocol
Time Frame: Data is available
Access Criteria: Email permission. Deidentified information only

REFERENCES:
- [Background] Gibran NS; Committee on Organization and Delivery of Burn Care, American Burn Association. Practice Guidelines for burn care, 2006. J Burn Care Res. 2006 Jul-Aug;27(4):437-8. doi: 10.1097/01.BCR.0000226084.26680.56. No abstract available. PMID 16819344
- [Background] Cuignet O, Pirson J, Soudon O, Zizi M. Effects of gabapentin on morphine consumption and pain in severely burned patients. Burns. 2007 Feb;33(1):81-6. doi: 10.1016/j.burns.2006.04.020. Epub 2006 Oct 30. PMID 17071002
- [Background] Summer GJ, Puntillo KA, Miaskowski C, Green PG, Levine JD. Burn injury pain: the continuing challenge. J Pain. 2007 Jul;8(7):533-48. doi: 10.1016/j.jpain.2007.02.426. Epub 2007 Apr 16. PMID 17434800
- [Background] Dierking G, Duedahl TH, Rasmussen ML, Fomsgaard JS, Moiniche S, Romsing J, Dahl JB. Effects of gabapentin on postoperative morphine consumption and pain after abdominal hysterectomy: a randomized, double-blind trial. Acta Anaesthesiol Scand. 2004 Mar;48(3):322-7. doi: 10.1111/j.0001-5172.2004.0329.x. PMID 14982565
- [Background] Gray P, Williams B, Cramond T. Successful use of gabapentin in acute pain management following burn injury: a case series. Pain Med. 2008 Apr;9(3):371-6. doi: 10.1111/j.1526-4637.2006.00149.x. PMID 18366516
- [Background] Dworkin RH. An overview of neuropathic pain: syndromes, symptoms, signs, and several mechanisms. Clin J Pain. 2002 Nov-Dec;18(6):343-9. doi: 10.1097/00002508-200211000-00001. PMID 12441827
- [Background] Dworkin RH, O'Connor AB, Backonja M, Farrar JT, Finnerup NB, Jensen TS, Kalso EA, Loeser JD, Miaskowski C, Nurmikko TJ, Portenoy RK, Rice ASC, Stacey BR, Treede RD, Turk DC, Wallace MS. Pharmacologic management of neuropathic pain: evidence-based recommendations. Pain. 2007 Dec 5;132(3):237-251. doi: 10.1016/j.pain.2007.08.033. Epub 2007 Oct 24. PMID 17920770

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 1/2010 to 9/13/2011. Patients were recruited for the study if they met criteria and were admitted for burn injuries.
Pre-assignment Details: There were no significant events or approaches following enrollment. Patients were randomized into groups.
Groups:
- Sugar Pill: Patients in this group received a sugar pill which looked identical to gabapentin.
- Gabapentin: Patients in this group received gabapentin which looked just like the sugar pill.
Period: Initial Study Period
Arm/Group | Sugar Pill | Gabapentin
Started | 26 | 27
Completed | 24 | 25
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Follow up
Arm/Group | Sugar Pill | Gabapentin
Started | 26 | 27
Completed | 19 | 24
Not Completed | 7 | 3
Not completed — Lost to Follow-up | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Gabapentin | Total
Number analyzed (Participants) | 26 | 27 | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 25 | 24 | 49
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (14.3) | 42.9 (11.6) | 41.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 24 | 23 | 47
Region of Enrollment [Number; unit: participants]
  United States | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Opioid Consumption Between the Treatment and the Control Groups (Morphine Equivalents)
Time Frame: From time of enrollment to 2 weeks after being discharged
Population: This was an intention to treate analysis. We measured the oral morphine equivalents both groups were administered.
Measure: Mean (Standard Deviation); unit: morphine equivalents
Groups:
- Placebo: Patients received a sugar pill similar to gabapentin.
- Gabapentin: Patients received gabapentin.
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 26 | 27
morphine equivalents | 7.0 (8.4) | 6.7 (11.6)
Statistical Analysis 1: Comparison: Placebo vs Gabapentin; Test type: Superiority; p < 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Gabapentin; Test type: Superiority; p < 0.04, Regression, Logistic

2. Secondary Outcome: Psychological Functioning as Evaluated by the Brief Symptom Inventory (BSI) Between Treatment and Placebo Groups
Description: The Brief Symptom Inventory 18 (BSI 18) is designed with reliability in mind. The BSI 18 assessment gathers patient-reported data to help measure psychological distress and psychiatric disorders in medical and community populations. As the latest in an integrated series of test instruments that include the SCL-90-R®, BSI® (53 questions), and DPRS® instruments, the BSI 18 test offers a more effective, easy-to-administer tool to help support clinical decision-making and monitor progress throughout treatment. BSI-18 measures three dimensions with 6 questions a piece (somatization , depression , anxiety) and overall psychological distress scores (Global severity index, GSI). Each of the 18 items range from a score of 0-4; total score ranges from 0-72 with higher scores indicating worse function. The GSI score is calculated as the mean of the three subscales. The study reported the GSI score. Higher score is worse.
Time Frame: First Clinic Follow Up After Discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 19 | 24
units on a scale | 9 (7.5) | 7.3 (7.2)
Statistical Analysis 1: Comparison: Placebo vs Gabapentin; Test type: Superiority; p < 0.8, t-test, 2 sided

3. Secondary Outcome: Difference in Psychological Outcomes on the Sickness Inventory Profile (SIP)
Description: The sickness inventory profile (SIP) is a behaviorally based measure of health status. Scores range from 0-68 with higher numbers indicating worse outcomes. The study report total SIP score. The higher the score the worse the function.
Time Frame: First Clinic Follow Up After Discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Gabapentin
Number analyzed (Participants) | 19 | 24
units on a scale | 34.9 (15.7) | 36.0 (19.5)
Statistical Analysis 1: Comparison: Placebo vs Gabapentin; Test type: Superiority; p = 0.8, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 0/26 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No